CLINICAL TRIAL: NCT06112730
Title: Nutritional Supplementation With Indirect Calorimetry During Pulmonary Rehabilitation in Patients With Chronic Respiratory Disease
Brief Title: Nutritional Supplementation in Patients With Chronic Respiratory Disease
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fu Jen Catholic University (Other)
Responsible Party: Principal Investigator, Ke-Yun, Chao, Group leader of Respiratory Therapists, Fu Jen Catholic University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: FJUH112271
Record Dates: First submitted 2023-10-29; First posted 2023-11-01 (Actual); Last update posted 2024-02-02 (Actual); Status verified 2024-02

CONDITIONS: Chronic Lung Disease
Keywords: Chronic obstructive pulmonary disease; Pulmonary rehabilitation; Nutritional supplementation; Indirect calorimetry
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard pulmonnary rehabilitation group (Active Comparator): Received routine pulmonnary rehabilitation
  Interventions: Other: Standard pulmonnary rehabilitation
- Nutritional supplementation intervention group (Experimental): Received regular pulmonnary rehabilitation plus healthy dietary recommendations
  Interventions: Other: Nutritional supplementation intervention

INTERVENTIONS:
Other: Standard pulmonnary rehabilitation — Undergo routine pulmonary rehabilitation without dietary intervention
  Arms: Standard pulmonnary rehabilitation group
Other: Nutritional supplementation intervention — Receive personalized dietary guidelines based on indirect calorimetry assessment
  Arms: Nutritional supplementation intervention group

SUMMARY:
The aim of this study is to investigate the nutritional status of patients with chronic pulmonary disease undergoing regular outpatient pulmonary rehabilitation.

DETAILED DESCRIPTION:
Background：

Exercise limitation due to impaired respiratory function is a common problem for COPD patients, and reduced muscle mass and malnutrition can exacerbate symptoms, impacting their functional ability and quality of life. Underweight COPD patients have an increased risk of mortality and acute exacerbations. Therefore, monitoring the body composition, nutritional status, and metabolic state of COPD patients and providing adequate nutritional support are crucial aspects of COPD management.Compared to healthy older adults, COPD patients require higher protein intake. Most studies have focused on analyzing body composition, respiratory and limb muscle strength, exercise performance, physical activity, lung function, emotional perception, and self-perceived scales, with limited assessment and exploration of calorie intake. Moreover, calorie intake estimation has mostly relied on formulas, lacking personalized and accurate assessment through indirect calorimetry.

Study Design：

This study is a single-center, prospective, randomized controlled trial.

Methods：

COPD patients who meet the inclusion criteria will be enrolled and randomly assigned to either the nutritional supplementation intervention group (experimental group) or the standard pulmonary rehabilitation group (control group). The experimental group will receive personalized dietary guidelines based on indirect calorimetry assessment by a nutritionist, while the control group will undergo routine pulmonary rehabilitation without dietary intervention. The study will follow up for a duration of 12 weeks, collecting data on cardiopulmonary physiological parameters, body composition, muscle strength, exercise performance, and indirect calorimetry assessment. Additionally, we will calculate the differences in recommended calorie intake between formula estimation and indirect calorimetry.

Effect：

We anticipate that indirect calorimetry will yield different results for calorie estimation compared to weight estimation and the Harris-Benedict equation. The nutritional supplementation intervention is expected to lead to improved changes in body composition, enhanced exercise performance and muscle strength, as well as better cardiopulmonary physiological parameters and self-perceived ratings.

Key words：

Chronic obstructive pulmonary disease, pulmonary rehabilitation, nutritional supplementation, indirect calorimetry

ELIGIBILITY:
Inclusion Criteria:

* Age between 45 and 80 years
* A written informed consent
* Pre-COPD or COPD stages I-IV as per the 2023 GOLD guidelines
* Recieved pulmonary rehabilitation at least three months
* Unwilling to nutritional outpatient assessment

Exclusion Criteria:

* Diagnosed with neuromuscular diseases
* Emergency room visits or hospitalizations for exacerbation of respiratory disease within three months
* Inability to cooperate with cardiopulmonary exercise testing
* Significant malnutrition or low BMI

Ages: 45 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2023-10-30 (Actual); Primary Completion 2024-06-30 (Estimated); Study Completion 2024-07-31 (Estimated)

PRIMARY OUTCOMES:
Resting energy expenditure | 15 minutes
  Basal metabolic rate

CONTACTS AND LOCATIONS:
Overall Officials: Ke-Yun Chao, PhD, Principal Investigator — Fu Jen Catholic University Hospital
Locations (1):
- Fu Jen Catholic University Hospital, Fu Jen Catholic University, New Taipei City, Taiwan

IPD SHARING:
Plan to Share IPD: No